CLINICAL TRIAL: NCT07015216
Title: Investigation of the Effects of Virtual Reality-Assisted Dual Task Training on Cerebral, Peripheral, and Respiratory Muscle Oxygenation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Virtual Reality-Assisted Dual Task Training on Muscle Oxygenation in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Berrak Varhan, Assistant Professor, PhD, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-02
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: Chronic Obstructive Lung Disease; dual task training; oxygenation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Conventional therapy + virtual reality-assisted dual task training
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Assisted Dual Task Training Group (Experimental): Virtual reality-based training will be conducted at ISÜFİZYOTEM in a custom-designed augmented VR environment. A 3D avatar and interactive scene (a 1 km crowded street) will be developed using Blender and Adobe Mixamo, with audio components from the Unity Asset Store. Participants will follow the avatar and perform exercises via a VR headset. After 1 minute of self-paced walking, a three-stage Stroop test will be introduced as a dual-task challenge. Sessions will be 20 minutes, supervised by a physiotherapist, with optional breaks. The intervention will be performed 3 times per week for 6 weeks.
  Interventions: Other: VR-Assisted Dual Task Training; Other: Conventional Therapy Program
- Conventional Therapy Program (Other): A pulmonary rehabilitation program will be administered to individuals with COPD once daily, three days per week for six weeks. The program will include diaphragmatic, chest, and bilateral segmental breathing exercises, breathing control training, relaxation positioning, peripheral muscle strengthening, and airway clearance techniques. Exercises will be explained and prescribed as a home-based program, to be performed twice daily with 10 repetitions. Patients will be given a daily log sheet to record adherence, which will be regularly monitored.
  Interventions: Other: Conventional Therapy Program

INTERVENTIONS:
Other: VR-Assisted Dual Task Training — Virtual reality-based training will be conducted at ISÜFİZYOTEM in a custom-designed augmented VR environment. A 3D avatar and interactive scene (a 1 km crowded street) will be developed using Blender and Adobe Mixamo, with audio components from the Unity Asset Store. Participants will follow the avatar and perform exercises via a VR headset. After 1 minute of self-paced walking, a three-stage Stroop test will be introduced as a dual-task challenge. Sessions will be 20 minutes, supervised by a physiotherapist, with optional breaks. The intervention will be performed 3 times per week for 6 weeks.
  Arms: VR-Assisted Dual Task Training Group
Other: Conventional Therapy Program — A pulmonary rehabilitation program will be administered to individuals with COPD once daily, three days per week for six weeks. The program will include diaphragmatic, chest, and bilateral segmental breathing exercises, breathing control training, relaxation positioning, peripheral muscle strengthening, and airway clearance techniques. Exercises will be explained and prescribed as a home-based program, to be performed twice daily with 10 repetitions. Patients will be given a daily log sheet to record adherence, which will be regularly monitored.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common but preventable disease that is associated with a chronic inflammatory response in the airways and lungs to noxious gases, often progressive, resulting in a persistent limitation of airflow. Chronic cough, dyspnea, and sputum production are the most common symptoms of the disease. Respiratory failure and decrease in physical activity seen in the later stages of the disease also negatively affect the participants' participation in daily life. COPD, which is an important health problem due to its increasing incidence, high prevalence, and associated social and economic costs, ranks fourth among the global causes of death.

Cognitive and physical impairments are often associated with COPD prognosis. In the literature, a relationship was found between prefrontal cortex activity, exercise tolerance, and dyspnea perception of the individual. The prevalence of cognitive impairment in COPD ranges from 10 to 61%. Considering the effect of cognitive function on motor control, it is thought to affect physical performance. Studies have reported that prefrontal cortex oxygenation and perfusion increase with exercise. Depending on the positive effect of neuron metabolism, increases in cognitive and physical functions are observed.

When examining the results of dual-task training and virtual reality applications in geriatric and neurological populations, positive effects on physical and cognitive functions have been demonstrated. Dual-task training causes an increase in cerebral perfusion and oxyhemoglobin as it requires more cognitive resources. Therefore, it is important for the investigators to create a program that includes cognitive performance rather than focusing only on motor performance in the rehabilitation of patients with COPD. Virtual reality applications are also widely used in many areas. A limited number of studies conducted on individuals with COPD have shown positive effects on physical performance. When examining the literature, it is seen that there is no study investigating the effects of virtual reality-assisted dual-task training in individuals with COPD.

Based on this information, the investigators aim to evaluate the effect of virtual reality-supported dual-task training on cerebral, peripheral muscle, and respiratory muscle oxygenation in individuals with COPD using the fNIRS imaging method. The 30 individuals with COPD included in the study will be divided into two groups as intervention and control groups. In addition to the conventional physiotherapy and rehabilitation program, virtual reality-supported dual-task training will be given to the intervention group. In the control group, only the conventional physiotherapy and rehabilitation program will be applied. The treatment program will continue for 6 weeks, 3 days a week in both groups. Within the scope of the project, respiratory muscle strength, respiratory function, peripheral muscle strength, fatigue, balance, functional capacity, activity of daily living, cognitive level, and cerebral, peripheral, and respiratory muscle oxygenation of both groups will be evaluated before and after the intervention, and the effects of the intervention will be examined.

For these purposes, the study will be the first in the literature to evaluate the effect of virtual reality-supported dual-task training in terms of cognitive functions and oxygenation and compare it with conventional physiotherapy applications.

The study results will provide a basis for determining an optimal non-pharmacological treatment method to protect and improve physical and cognitive performance in individuals with COPD. In addition, the investigators believe that the study will have a social impact by helping to reduce mortality and morbidity rates in these patients and indirectly alleviate the burden on healthcare services. This project will contribute to the literature by providing a different perspective for clinical applications, as well as serving as a guide for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD stage 2 or 3 according to GOLD classification
* No orthopedic and/or neuromuscular conditions that would interfere with dual-task training
* Ability to ambulate
* Adequate cognitive level to participate in the training (Mini Mental State Examination score ≥ 23)
* Voluntary participation

Exclusion Criteria:

* Presence of vestibular problems that would interfere with virtual reality applications
* Visual impairments
* Any medical condition contraindicating exercise participation
* Being in an acute exacerbation period
* Having an active infection
* Diagnosis of cancer
* Known cardiovascular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-12 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake (VO₂max) | Baseline and after 6 weeks of intervention
  Maximal oxygen consumption (VO₂max) will be measured during incremental cardiopulmonary exercise testing (CPET) using a COSMED metabolic system and cycle ergometer. VO₂max is defined as the highest oxygen uptake achieved during the final stage of exercise.
Cognitive Function (MoCA Score) | Baseline and after 6 weeks of intervention
  Cognitive status will be assessed using the Montreal Cognitive Assessment (MoCA). Scores range from 0 to 30, with lower scores indicating more severe impairment.
Dual Task Effect on Gait Speed (DTE %) | Baseline and after 6 weeks of intervention
  The effect of performing a cognitive task while walking will be quantified as the percentage change in gait speed compared to normal walking.
Cortical Activation During Dual Tasks - Oxyhemoglobin (O₂Hb) | Baseline and after 6 weeks of interventio
  Functional near-infrared spectroscopy (fNIRS) will be used to measure changes in cortical oxyhemoglobin (O₂Hb) levels during dual task performance, indicating increased neural activation.
Cortical Activation During Dual Tasks - Deoxyhemoglobin (HHb) | Baseline and after 6 weeks of intervention
  Functional near-infrared spectroscopy (fNIRS) will be used to measure changes in cortical deoxyhemoglobin (HHb) levels during dual task performance, reflecting changes in oxygen consumption and blood flow.

SECONDARY OUTCOMES:
Dyspnea Severity | Pre- and post-intervention (6 weeks).
  Self-reported scale ranging from 0-4 to assess dyspnea level.
Fatigue Severity | Pre- and post-intervention (6 weeks).
  9-item scale to assess fatigue over the past month; each item rated 1-7.
Maximal Inspiratory Pressure (MIP) | Pre- and post-intervention (6 weeks)
  MIP will be measured using the Powerbreathe Plus MR device in accordance with ATS/ERS recommendations. This test assesses inspiratory muscle strength.
Maximal Expiratory Pressure (MEP) | Pre- and post-intervention (6 weeks)
  MEP will be measured using the Powerbreathe Plus MR device in accordance with ATS/ERS recommendations. This test assesses expiratory muscle strength.
Forced Expiratory Volume in 1 Second (FEV₁) | Pre- and post-intervention (6 weeks)
  FEV₁ will be measured using the Cosmed Pony FX spirometer according to ATS/ERS guidelines. This parameter reflects airway obstruction.
Forced Vital Capacity (FVC) | Pre- and post-intervention (6 weeks)
  FVC will be measured using the Cosmed Pony FX spirometer in accordance with ATS/ERS standards. It represents the total volume of air exhaled during a forced breath.
FEV₁/FVC Ratio | Pre- and post-intervention (6 weeks)
  The ratio of FEV₁ to FVC will be calculated to evaluate airflow limitation. Measurements will be taken using the Cosmed Pony FX spirometer per ATS/ERS guidelines.
Peak Expiratory Flow (PEF) | Pre- and post-intervention (6 weeks)
  PEF will be measured using the Cosmed Pony FX spirometer, following ATS/ERS guidelines. It indicates the highest flow achieved during a forced exhalation.
Forced Expiratory Flow 25-75% (FEF₂₅-₇₅) | Pre- and post-intervention (6 weeks)
  FEF₂₅-₇₅ will be measured using the Cosmed Pony FX spirometer to assess the flow during the middle half of the forced vital capacity. Measurements follow ATS/ERS standards.
Carbon Monoxide Level (Smokerlyzer Device) | Pre- and post-intervention (6 weeks).
  Non-invasive CO level measurement.
Daily Living Activities | Pre- and post-intervention (6 weeks).
  (London Chest Activity of Daily Living Scale - LCADL) 15 items scored 0-5 assessing dyspnea in daily tasks.
Hand Grip Strength | Pre- and post-intervention (6 weeks).
  Three repeated trials with best score recorded.
Flamingo Balance Test | Pre- and post-intervention (6 weeks)
  The Flamingo Balance Test assesses static balance by measuring the ability to maintain a single-leg stance. The participant stands on one leg on a narrow beam, and the number of balance losses (falls) in 60 seconds is recorded. Fewer falls indicate better balance.
Functional Reach Test (FRT) | Pre- and post-intervention (6 weeks)
  The Functional Reach Test evaluates dynamic balance by measuring how far a person can reach forward beyond arm's length while maintaining a fixed base of support in standing. The reach distance in centimeters is recorded; longer reach indicates better dynamic balance.
Heart Rate Monitoring | Pre- and post-intervention, and during CPET recovery (1, 3, 5 minutes)
  Heart rate (HR) will be measured in beats per minute (bpm) using a pulse oximeter or electrocardiogram. Values will be recorded at rest (pre- and post-intervention) and during recovery following cardiopulmonary exercise testing (CPET) at 1, 3, and 5 minutes.
Blood Pressure Measurement | Pre- and post-intervention, and during CPET recovery (1, 3, 5 minutes
  Systolic and diastolic blood pressure (SBP/DBP) will be measured in mmHg using a standard sphygmomanometer or automated blood pressure device. Measurements will be taken at rest (pre- and post-intervention) and during CPET recovery at 1, 3, and 5 minutes.
Peripheral Oxygen Saturation (SpO₂) | Pre- and post-intervention, and during CPET recovery (1, 3, 5 minutes)
  SpO₂ will be measured using a fingertip pulse oximeter. Values will be recorded as a percentage (%) at rest (pre- and post-intervention) and during CPET recovery at 1, 3, and 5 minutes.
Respiratory Rate Monitoring | Pre- and post-intervention, and during CPET recovery (1, 3, 5 minutes)
  Respiratory rate (breaths per minute) will be measured by manual observation or via monitoring device. Data will be collected at rest (pre- and post-intervention) and at 1, 3, and 5 minutes during CPET recovery.
Peripheral Muscle Strength Assessment Using Medical Research Council (MRC) Scale | Pre- and post-intervention (6 weeks)
  Peripheral muscle strength will be evaluated using the Medical Research Council (MRC) scale. This semi-quantitative scale grades muscle strength from 0 (no contraction) to 5 (normal strength) across selected muscle groups, including upper and lower extremities. The total MRC sum score provides an estimate of global muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Istınye University, Istanbul,, Istanbul, Turkey (Türkiye)